CLINICAL TRIAL: NCT05892224
Title: Research on Brain Function of Metabolism-based Artificial Intelligence Assisted Clinical Classification of Obesity
Brief Title: Study on Brain Function of Obesity Classification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Qu, Clinical Professor and Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: Brain function in obesity
Record Dates: First submitted 2023-03-10; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Functional Neuroimaging
Keywords: obesity; Functional Neuroimaging; Brain; artificial intelligence
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- MHO group: Metabolic healthy obesity
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- HMO-U group: Hypermetabolic obesity-hyperuricemia
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- HMO-I group: Hypermetabolic obesity-hyperinsulinemia
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- LMO group: Hypometabolic obesity
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- control group: Healthy person

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Obese patients of different subtypes were all expected to undergo bariatric surgery
  Groups: HMO-I group; HMO-U group; LMO group; MHO group

SUMMARY:
The purpose of this study was to investigate the differences and similarities of brain function in patients with four subtypes of obesity, and the relationship between brain function changes and complications after weight loss and metabolic improvement. 120 patients with obesity and 30 healthy individuals with normal BMI were enrolled.

DETAILED DESCRIPTION:
Although the investigators have clinically observed significant differences in appetite and metabolic status in patients with the above four types of obesity, the brain functional characteristics of different obesity subtypes and their relationship with metabolic markers are still unclear. Based on this, in this project, the investigators plan to explore further the similarities and differences in brain function in patients with four subtypes of obesity and the relationship between brain function changes after weight loss and metabolic improvement and the occurrence of complications.

120 patients with obesity and 30 healthy individuals with normal BMI were enrolled.

All patients with obesity underwent LSG. A multidisciplinary team evaluated participants with obesity at baseline, 1, 3, 6, and 12 months after laparoscopic sleeve gastrectomy (LSG). Anthropometrics, Metabolic indicators, sex hormones, menstruation，glucose-lipid metabolic markers, and hepatic steatosis assessed by FibroScan(CAP value and E value) were measured baseline and postoperative. Resting and task state functional magnetic resonance imaging (fMRI) measurements were performed at baseline for all participants at two-time points before and after meals. Measurements were repeated in obese patients 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 16-65 years old
* BMI over 37.5kg/m2, or BMI over 32.5kg/m2 with diabetes which meets the recommended cut-off bariatric surgery of the Guidelines for surgical treatment of obesity accompanied with or without type 2 diabetes in China.

Exclusion Criteria:

* secondary causes of obesity such as hypothalamic obesity, Cushing syndrome, hypophysis dysfunction, etc
* pregnancy or location
* contraindications for laparoscopic surgery, such as gastrointestinal diseases of intra-abdominal infection, adhesion, etc
* severe heart, liver, and kidney dysfunction
* organic and systemic diseases intolerant of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 Patients from Shanghai Tenth People's Hospital were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging of brain | 6 months
  The subjects underwent fMRI scans before and after eating. Blood oxygen levels depend on functional brain imaging (Blod-fMRI) to collect the brain's local BLOD response (hemodynamic response) caused by the electrical activity of neurons. The stronger the BLOD response, the more excitability of the local brain.
  A region-of-interest (ROI) approach was applied with the use of masks that were established in an independent study of normal-weight subjects to be markers of satiety or predictors of food choices. ROIs included the left and right ventral striatum (nucleus accumbens), the left and right amygdala, the left and right dorsal striatum (caudate and putamen), the left and right insula, and the medial orbital frontal cortex (mOFC).
  functional connectivity analysis analyzes the compatibity of temporal signals of two or more pairs of brain regions or the differences in the strength of functional connections under different experimental conditions

SECONDARY OUTCOMES:
BMI | 12 months
  BMI=weight(kg)/height(m)^2
Waist/hip Ratio | 12 months
  WHR(waist-hip ratio)=Waist Circumference in centimeter/Hip Circumference in centimeter
DXA(dual energy x-ray absorptiometry) | 12 months
  Dual X-ray Absorptiometry body composition analysis
Abdominal Fat Measurement | 12 months
  Abdominal Fat Measurement by B-mode Ultrasound
FBG | 12 months
  fasting blood-glucose in mmol/L
PBG | 12 months
  postprandial blood-glucose in mmol/L
FINS | 12 months
  fasting serum insulin in mU/L
PINS | 12 months
  postprandial insulin in mU/L
ALT | 12 months
  alanine aminotransferase in U/L
AST | 12 months
  aspartate aminotransferase in U/L
UA | 12 months
  Uric acid in umol/L
HOMA-IR | 12 months
  Homeostatic model assessment insulin resistance index=FBG*FINS/22.5
HbA1c (%) | 12 months
  Glycated hemoglobin
LDL-C | 12 months
  low-density lipoprotein cholesterol in mmol/L
HDL-C | 12 months
  Hight-density lipoprotein cholesterol in mmol/L
TT | 12 months
  total testosterone in nmol/L
SHBG | 12 months
  sex hormone-binding globulin in nmol/L
TSH | 12 months
  thyroid stimulating hormone in μIU/ml
FT3 | 12 months
  free triiodothyronine in pmol/L
FT4 | 12 months
  free thyroxine in pmol/L
FT | 12 months
  free testosterone (nmol/L)
DHEAS | 12 months
  Dehydroepiandrosterone Sulfate (ug/dl)
PTH | 12 months
  parathyroid hormone in （ng ／ L）
25OHD | 12 months
  25 hydroxyvitamin D in （nmol ／ L）
Ca | 12 months
  serum calcium in (mmol/L)
GLP-1 | 12 months
  Glucagon-like peptide-1(pmol/L)
LCN2 | 12 months
  Lipocalin 2 level
Ghrelin | 12 months
  Ghrelin level
Leptin | 12 months
  Leptin level
S100 | 12 months
  S100 protein level
GFAP | 12 months
  Glial fibrillary acidic protein level
TEFQ-R21 | 12 months
  The TFEQ-R21 consisted of 21 items rated on a four-point Likert scale. We averaged the scores (ranging from 1 to 4) for the overall items as well as the items within the subdomain of each item, i.e., EE, UE, and CR, where a higher score indicated a more dysfunctional eating behavior.
HADS | 12 months
  HADS consists of two subscales: HADS-A, designed to detect anxious states, and HADS-D, designed to detect depressive states. Each subscale consists of seven items with a 4-point ordinal response format. Scores ranges from 0 to 21 in each subscale, with higher scores indicating higher levels of anxious or depressive state. Participants answer each item thinking of how they felt and/or behaved during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr., Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No